CLINICAL TRIAL: NCT06560697
Title: Randomized Phase II Study to Measure the Safety and Efficacy of Concomitant CT/RT Followed by Ablative Stereotactic Radiotherapy (SABR) vs Brachytherapy in Patients With Cervical Carcinoma in Clinical Stage IB3-IIIC1 at INCAN
Brief Title: Cervical Boost by Ablative Stereotactic Radiotherapy (SABR) vs Brachytherapy in Patients With Cervical Carcinoma
Acronym: SABRVICAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cancerología (Other Government)
Collaborators: National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (023/044/ICI) (CEI/016/23)
Record Dates: First submitted 2024-07-19; First posted 2024-08-19 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Uterine Cervical Neoplasm
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized open-label phase 2 study in people with CaCu clinical stages IB3-IIIC1 treated with QT/RT. Subjects will be randomized to cervical boost with SBRT or 3D intracavitary brachytherapy in a 1:1 ratio and stratified by nodal status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cervical Boost with SABR (Experimental): patients with CC clinical stages IB3-IIIC1 who will be treated with CT/RT with a minimum dose of 45Gy and boost in the case of macroscopic nodes (1.8Gy per fraction from Monday to Friday) with cisplatin and cervical boost with SBRT of 28Gy in 4 fractions administered at least every 40 hours to achieve an EQD210(Gy) at PTV D90% of 83.9Gy
  Interventions: Radiation: SABR VS Intracavitary 3D Brachytherapy
- Cervical Boost with Intracavitary Brachytherapy (Active Comparator): Patients with CC clinical stages IB3-IIIC1 will be treated with CT/RT with a minimum dose of 45Gy and boost in the case of macroscopic nodes (1.8Gy per fraction from Monday to Friday) with cisplatin and cervical boost with high-dose-rate 3D brachytherapy with a dose of 28Gy in 4 fractions administered at least every 40 hours to achieve an EQD210(Gy) at point A of 83.9Gy.
  Interventions: Radiation: SABR VS Intracavitary 3D Brachytherapy

INTERVENTIONS:
Radiation: SABR VS Intracavitary 3D Brachytherapy — Arm 1 will be the experimental arm and will consist of patients with CC clinical stages IB3-IIIC1 who will be treated with CT/RT with a minimum dose of 45Gy and boost in the case of macroscopic nodes (1.8Gy per fraction from Monday to Friday) with cisplatin and cervical boost with SBRT of 28Gy in 4 fractions administered at least every 40 hours to achieve an EQD210(Gy) at PTV D90% of 83.9Gy. Arm 2 will be the control arm that will consist of patients with CC clinical stages IB3-IIIC1 and will be treated with CT/RT with a minimum dose of 45Gy and boost in the case of macroscopic nodes (1.8Gy per fraction from Monday to Friday) with cisplatin and cervical boost with high-dose-rate 3D brachytherapy with a dose of 28Gy in 4 fractions administered at least every 40 hours to achieve an EQD210(Gy) at point A of 83.9Gy.

SUMMARY:
Background Cervical cancer (CaCu) is the fourth cause of death in women. In patients with locally advanced disease, the treatment of choice is CT/RT, followed by additional boosting with brachytherapy (BT). There is an international decrease in the use of this technique due to financial restrictions. Given the difficulties in using brachytherapy as a boost, several series have described promising results in local control using boost with highly conformal techniques such as stereotactic body radiotherapy (SBRT). On the other hand, prospective studies are scarce and with controversial results. No study has been published that directly compares three-dimensional intracavitary SBRT and BT. In this clinical trial, the researchers aim to demonstrate that boosting with SBRT is not inferior to intracavitary brachytherapy in patients with CC.

Methodology

Primary Objective:

To evaluate the safety and efficacy of concomitant CT/RT followed by Ablative Body Stereotactic Radiotherapy (SBRT) vs Brachytherapy in patients with Cervical Cancer in clinical stage IB3-IIIC1 at INCan.

Secondary Objectives:

The purpose of this study is to evaluate quality of life, local efficacy (local control and time to local recurrence), overall survival, disease-free survival, and time to distant recurrence.

Study Design:

SABRVICAL is a meticulously designed randomized two-arm open-label phase II study to compare QT/RT + SBRT vs QT/RT + Brachytherapy. It will include patients with IB3-IIIC1 CaCu >18 years of age with adequate renal function. They will be randomized 1:1 to the experimental arm or the standard arm.

Expected Results and Outlook With this study, we aim to assess that the safety and efficacy of concomitant QT/RT with cisplatin followed by SBRT is not inferior to boost with brachytherapy in patients with CaCu IB3-IIIC1. The potential impact of this study is significant, as it could provide new treatment options for hospitals that do not have brachytherapy or have a prolonged waiting list for this procedure.

DETAILED DESCRIPTION:
A randomized phase 2 trial is required for two reasons:

1. The literature lacks enough prospective information. In this context, a randomized phase 2 study would identify SBRT as a promising experimental treatment that, depending on the results, could be tested in a phase 3 trial.
2. Randomization will provide an adequate control group to serve as a comparator for the experimental arm since non-randomized historical or contemporary controls are not appropriate due to the amount of bias they introduce in patient selection as well as confounders (use of 2D brachytherapy). instead of 3D or the use of conformal radiotherapy and not intensity-modulated radiotherapy).

To evaluate the safety and efficacy of concomitant CT/RT followed by SBRT vs high rate 3D Intracavity Brachytherapy in patients with Cervical Cancer in clinical stage IB3-IIIC1 at INCan:

1. Evaluate the safety of CT/RT using the CTCAE V5.0 criteria.
2. Evaluate local efficacy and objective response using the RECIST 1.1 criteria.
3. Compare the time to local, regional, and distant recurrence between radiotherapy techniques.
4. Compare overall survival and progression-free survival between both radiotherapy techniques.
5. Measure the patient's quality of life using the QLQ-C30 and QLQ-CX24 questionnaires.

Randomized open-label phase 2 study in people with CaCu clinical stages IB3-IIIC1 treated with QT/RT. Subjects will be randomized to cervical boost with SBRT or 3D intracavitary brachytherapy in a 1:1 ratio and stratified by nodal status.

Arm 1 will be the experimental arm and will consist of patients with CC clinical stages IB3-IIIC1 who will be treated with CT/RT with a minimum dose of 45Gy and boost in the case of macroscopic nodes (1.8Gy per fraction from Monday to Friday) with cisplatin and cervical boost with SBRT of 28Gy in 4 fractions administered at least every 40 hours to achieve an EQD210(Gy) at PTV D90% of 83.9Gy. Arm 2 will be the control arm that will consist of patients with CC clinical stages IB3-IIIC1 and will be treated with CT/RT with a minimum dose of 45Gy and boost in the case of macroscopic nodes (1.8Gy per fraction from Monday to Friday) with cisplatin and cervical boost with high-dose-rate 3D brachytherapy with a dose of 28Gy in 4 fractions administered at least every 40 hours to achieve an EQD210(Gy) at point A of 83.9Gy.

Sample size The maximum acceptable toxicity (grade 3 or higher) is 24%. The only phase II clinical trial published in the literature about SBRT in CC reported late toxicity of 26.7% at 2 years. For intracavitary brachytherapy, a grade 3 late toxicity of 3.31% has been reported.

The sample size was calculated using a formula for 2 proportions, in which an incidence of grade 3-4 toxicity of 26.7% for arm A and 3.31% for group B was considered. A α error of 5% and a power of 80%. A total of 35 patients for each arm are needed plus a 20% loss = 42 patients for each arm (see figure attached).

Inclusion criteria

1. People with cervical cancer >18 years of age.
2. Signed informed consent form approved by the regulatory committees of both institutes and, obtained before each procedure related to the protocol, and that is not considered part of the normal care of the patient.
3. Able to comply with scheduled visits, treatment schedules, laboratory and imaging studies, and completing quality of life questionnaires.
4. Histological confirmation of CaCu and staged as IB3-IIIC1.
5. Squamous cell, adenosquamous, or adenocarcinoma histology.
6. No prior treatment for cervical cancer.
7. With disease measurable by CT, MRI, or PET/CT according to REC 1.1 criteria. This measurement must be carried out 28 days before randomization.
8. Functional status of 0-2 according to WHO criteria.
9. Charlson Comorbidity Index of 1-4
10. Candidates to receive cisplatin.
11. Normal hematological, kidney, and hepatic function according to:

    Hematological:

    Hemoglobin equal to or >10g/L. (With the possibility of transfusion prior to treatment to reach this hemoglobin level).

    Leukocytes >4000/mm3. Platelets>100,000mm3. Neutrophils >1500 / μL

    Hepatic:

    Total bilirubin <1.5 X times the normal value. Transaminases <1.5 X times the normal value.

    Renal:

    Creatinine <1.3mg/dl or creatinine clearance > 40 mL/minute (using the Cockcroft/Gault formula).

    Women: DepCr = (140 - Age in years) x Weight in kg x 0.85

    ___________________________________ 72 x Serum Creatinine in mg/dL Men: DepCr = (140 - Age in years) x Weight in kg x 1.00

    _____________________________________ 72 x Serum Creatinine in mg/dL
12. Chest tomography without metastatic disease or infectious diseases.
13. Negative pregnancy test in women of childbearing age.
14. Not a candidate for another clinical trial within the institution.

Exclusion Criteria

1. Patients with small-cell carcinoma or other rare histologies (glassy cell carcinoma, melanoma, sarcomas, lymphomas)
2. Patients with non-measurable disease.
3. Patients in whom pregnancy is confirmed during the recruitment procedure.
4. Clinical stages IIIC2-IVB.
5. Serious infections or diseases that can be reactivated with the use of chemotherapy or that could limit its use (hepatitis or HIV).
6. Pre-existing neuropathy of any etiology.
7. Concomitant treatment with another experimental drug.
8. Mental illnesses: With the intention of maximizing adherence to the study, those patients who are at risk of imminent physical aggression (evident during the interview), have intellectual disabilities or autism, and who come for consultation due to coercion will not be included in the study. their accompanying Severe major depressive disorder, with or without psychotic symptoms; patients in whom a psychiatric diagnosis coexists in addition to the abuse of some recreational substance, eating disorders, schizophrenia, or Bipolar-type Schizoaffective Disorder.
9. Grade 3 obesity with body mass index >40kg/m2 according to the World Health Organization: Patients treated with pelvic radiotherapy and a body mass index >40kg/m2 are associated with a decrease in quality of life due to sexual, intestinal, genitourinary alterations, as well as greater toxicity due to oncological treatments offered such as intracavitary brachyter in which the positioning of the equipment in the vaginal area is significantly difficult in sedated patients. Patients with grade III obesity will not be included.
10. Any patient who is absent from follow-up for 5 subsequent appointments will be excluded from the study.
11. History of total or partial hysterectomy.
12. Patients with a history of neoadjuvant chemotherapy or use of another antineoplastic drug differ from cisplatin (40 mg/m2).
13. History of use of Bevacizumab to manage a pathology other than CC or intention to use this drug as part of the treatment of CC.

15. Charlson Comorbidity Index >5 16. Synchronous Cancer except non-melanoma Skin Cancer. 17. History of pelvic irradiation for metachronous cancer. 18. Inflammatory bowel disease or collagen diseases. 19. Patients with severe immunosuppression (transplant or treatment with immunosuppressive drugs).

20. Patients who do not sign the informed consent form. 21. Suspected alcohol or recreational drug abuse. 22. Participation in any other clinical trial in the last 90 days prior to protocol recruitment.

23. Any illness or disability not covered by the exclusion criteria that, in the researchers' opinion, may put the patient's safety and compliance with the protocol at risk.

24. Patients with a percentage of rectal circumference receiving a dose of 15Gy >62.7%.

Elimination Criteria

A patient will be removed from the study for the following reasons:

1. If the patient requests it.
2. Inappropriate inclusion in the study without following the inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. People with cervical cancer >18 years of age.
2. Signed informed consent form approved by the regulatory committees of both institutes and, obtained before each procedure related to the protocol, and that is not considered part of the normal care of the patient.
3. Able to comply with scheduled visits, treatment schedules, laboratory and imaging studies, and completing quality of life questionnaires.
4. Histological confirmation of CaCu and staged as IB3-IIIC1.
5. Squamous cell, adenosquamous, or adenocarcinoma histology.
6. No prior treatment for cervical cancer.
7. With disease measurable by CT, MRI, or PET/CT according to REC 1.1 criteria. This measurement must be carried out 28 days before randomization.
8. Functional status of 0-2 according to WHO criteria.
9. Charlson Comorbidity Index of 1-4
10. Candidates to receive cisplatin.
11. Normal hematological, kidney, and hepatic function according to:

    Hematological:

    Hemoglobin equal to or >10g/L. (With the possibility of transfusion prior to treatment to reach this hemoglobin level).

    Leukocytes >4000/mm3. Platelets>100,000mm3. Neutrophils >1500 / μL

    Hepatic:

    Total bilirubin <1.5 X times the normal value. Transaminases <1.5 X times the normal value.

    Renal:

    Creatinine <1.3mg/dl or creatinine clearance > 40 mL/minute (using the Cockcroft/Gault formula).

    Women: DepCr = (140 - Age in years) x Weight in kg x 0.85

    ___________________________________ 72 x Serum Creatinine in mg/dL Men: DepCr = (140 - Age in years) x Weight in kg x 1.00

    _____________________________________ 72 x Serum Creatinine in mg/dL
12. Chest tomography without metastatic disease or infectious diseases.
13. Negative pregnancy test in women of childbearing age.
14. Not a candidate for another clinical trial within the institution.

Exclusion Criteria:

1. Patients with small-cell carcinoma or other rare histologies (glassy cell carcinoma, melanoma, sarcomas, lymphomas)
2. Patients with non-measurable disease.
3. Patients in whom pregnancy is confirmed during the recruitment procedure.
4. Clinical stages IIIC2-IVB.
5. Serious infections or diseases that can be reactivated with the use of chemotherapy or that could limit its use (hepatitis or HIV).
6. Pre-existing neuropathy of any etiology.
7. Concomitant treatment with another experimental drug.
8. Mental illnesses: With the intention of maximizing adherence to the study, those patients who are at risk of imminent physical aggression (evident during the interview), have intellectual disabilities or autism, and who come for consultation due to coercion will not be included in the study. their accompanying Severe major depressive disorder, with or without psychotic symptoms; patients in whom a psychiatric diagnosis coexists in addition to the abuse of some recreational substance, eating disorders, schizophrenia, or Bipolar-type Schizoaffective Disorder.
9. Grade 3 obesity with body mass index >40kg/m2 according to the World Health Organization: Patients treated with pelvic radiotherapy and a body mass index >40kg/m2 are associated with a decrease in quality of life due to sexual, intestinal, genitourinary alterations, as well as greater toxicity due to oncological treatments offered such as intracavitary brachyter in which the positioning of the equipment in the vaginal area is significantly difficult in sedated patients. Patients with grade III obesity will not be included.
10. Any patient who is absent from follow-up for 5 subsequent appointments will be excluded from the study.
11. History of total or partial hysterectomy.
12. Patients with a history of neoadjuvant chemotherapy or use of another antineoplastic drug differ from cisplatin (40 mg/m2).
13. History of use of Bevacizumab to manage a pathology other than CC or intention to use this drug as part of the treatment of CC.

15. Charlson Comorbidity Index >5 16. Synchronous Cancer except non-melanoma Skin Cancer. 17. History of pelvic irradiation for metachronous cancer. 18. Inflammatory bowel disease or collagen diseases. 19. Patients with severe immunosuppression (transplant or treatment with immunosuppressive drugs).

20. Patients who do not sign the informed consent form. 21. Suspected alcohol or recreational drug abuse. 22. Participation in any other clinical trial in the last 90 days prior to protocol recruitment.

23. Any illness or disability not covered by the exclusion criteria that, in the researchers' opinion, may put the patient's safety and compliance with the protocol at risk.

24. Patients with a percentage of rectal circumference receiving a dose of 15Gy >62.7%

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — People with uterine cervix carcinoma
Enrollment: 84 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute Toxicity | 5 years
  It will be measured using the CTCAE V5.0 criteria.
Chronic Toxicity | 5 years
  It will be measured using the CTCAE V5.0 criteria.

SECONDARY OUTCOMES:
General Health Perception | 5 years
  Quality of Life measured with the QLQ-C30 and QLQ-CX24 questionnaires validated in Mexican patients.
Local Control | 5 years
  Local efficacy and objective response using the RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, Tlalpan, Mexico